CLINICAL TRIAL: NCT07278505
Title: Pathophysiological Mechanisms of Cannabidiol in Stress Regulation
Brief Title: Study of Cannabidiol and Neuroimaging on Stress
Acronym: SCANS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Jazz Pharmaceuticals (Industry); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Keren Bachi, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STUDY-25-00337; 1R01MH139940 (NIH)
Record Dates: First submitted 2025-12-03; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Early Life Adversity; Trauma; Stress
Keywords: Cannabidiol; Childhood Trauma; Stress; Trauma; Anxiety; Adversity
MeSH Terms: conditions — Wounds and Injuries; Anxiety Disorders | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol (CBD) (Experimental): Cannabidiol - oral CBD solution 400 mg
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Drug: Placebo Inactive oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — 400mg cannabidiol
  Other Names: CBD; Epidiolex
  Arms: Cannabidiol (CBD)
Drug: Placebo — Inactive oral solution
  Arms: Placebo

SUMMARY:
Dysregulation in stress responsivity is a growing psychiatry-transdiagnostic fundamental phenomenon, with limited therapeutic strategies. With the legalization of medical and recreational cannabis, many people consume cannabidiol (CBD; a nonintoxicating cannabinoid) to alleviate stress response, without the benefit of scientific guidance. To address this gap, the investigators propose a rigorous translational neuroscience study in a clinical high-risk population to define the roles of CBD in stress response with mechanisms of mesocorticolimbic-network function and hierarchy, neurometabolic, endocrine, and behavior, building upon convergent evidence from animal models and human evidence from our laboratories.

DETAILED DESCRIPTION:
Dysregulation in stress responsivity, encompassing mesocorticolimbic and hypothalamus-pituitary-adrenal-axis pathways, is a psychiatry-transdiagnostic fundamental phenomenon. Current anxiolytic pharmacotherapies are limited in their efficacy and could cause dependence, low tolerance, and sexual dysfunction. With the growing number of vulnerable individuals suffering from stress-related disorders in society, there is an urgent need for novel therapeutic modalities particularly for early intervention and to improve treatments of stress-related disorders. Convergent evidence from animal and human studies of cannabidiol (CBD), a nonintoxicating and well-tolerated cannabinoid, has shown to have anxiolytic effects on stress reactivity especially in responses to environmental stimuli (cue-sensitized states). CBD has multiple pharmacological targets acting as an allosteric modulator of cannabinoid receptors and a glutamate-modulating agent. Despite recent surges in the use of CBD to alleviate stress symptoms, its pathophysiological mechanisms in human stress-system pathways remain largely unknown. Understanding the mechanisms of action of CBD in stress responsivity may lead to novel therapeutic strategies for stress-related disorders. Based on its safety and the growing evidence of CBD to reduce cue-induced reactivity, the investigators propose to evaluate the mechanisms underlying CBD's roles in stress response in a clinical high-risk population of young adults with early life adversity (ELA), known to exhibit this phenotype. This proposal leverages the investigators clinical and research expertise with high-risk populations with ELA and other investigators established experience with CBD clinical trials. Specifically, the researchers neuroimaging study demonstrated prefrontal neuroanatomical impairments associated with enhanced clinical symptomatology in individuals with ELA. In relation to CBD, the researchers have shown in healthy individuals that oral CBD is safe and well tolerated. The researchers have demonstrated that CBD reduced cue-induced anxiety in individuals with psychopathology and that the effects persisted even when the cannabinoid was no longer detectable in the body. Moreover, in the randomized, double-blind placebo-controlled trial the researchers not only replicated the original findings that CBD decreased cue-induced anxiety but also showed that it concomitantly reduced physiological stress responsivity marks (cortisol and heart rate). Importantly, its protracted effects were again evident a week after the last administration. Notably, the researchers pharmacokinetic trial replicated the previous findings showing rapid bioavailability in oral CBD dose (400mg) known to have behavioral efficacy. The investigators hypotheses are that during stress responsivity CBD will: 1) downregulate the neural reactivity in mesocorticolimbic regions; 2) reduce influence of limbic regions within the stress network dependency hierarchy; 3) reduce neuronal viability in mesocorticolimbic regions; and 4) decrease endocrine and behavioral hyperreactivity, in clinical high-risk individuals. This study of unmedicated young adult males and females (N=160) with ELA, will examine neurobiological mechanisms of stress as manipulated by acute CBD vs. placebo (400mg, oral; using a double-blind, randomized, placebo-control design), as well as determine the relationship between CBD-sustained (7-day) change and endocrine and behavioral acute stress responsivity.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and give informed consent.
* Individuals between 18 and 25 years old; Sex is used a biological factor (50% of individuals recruited will be females, allowing sex comparisons).
* English speakers.
* Cognitive performance at threshold of greater than or equal to 23 as assessed by the Montreal Cognitive Assessment (MoCA).
* Presence of ELA at threshold of at least one type of maltreatment measured by the Maltreatment and Abuse Chronology of Exposure (MACE) Scale and/or one type of maltreatment scored moderate/severe as measured by the Childhood Trauma Questionnaire (CTQ)
* Presence of moderate/heightened stress as measured with a score of greater than or equal to 14 on the Perceived Stress Scale and/or high trait anxiety at threshold score of greater than or equal to 40 as measured with the State-Trait Anxiety Inventory (STAI) and no greater than moderate anxiety scores (max. 14) as measured by the Generalized Anxiety Disorder-7 (GAD7)

Exclusion Criteria:

* Have a medical condition that would make study participation unsafe, and/or which would make treatment compliance difficult, and/or would prevent adherence to study procedure. This includes but is not limited to the following criteria: history of cardiac disease, arrhythmias, neurological disease of central origin, head trauma, and seizures.
* Meet criteria for any current psychiatric diagnosis as per DSM-5 [determined with the Mini International Neuropsychiatric Interview for DSM-5 (M.I.N.I. version 7.2)].
* Using any psychoactive drug (other than nicotine and/or alcohol) in the past seven days (determined by lack of acute withdrawal symptoms, the negative result of a urine drug screen, timeline follow back, and alcohol breathalyzer to detect alcohol intoxication).
* Positive urine drug screen (tetrahydrocannabinol, cocaine, opiates, benzodiazepines, barbiturates, amphetamines, morphine, methadone, methamphetamines, oxycodone, phencyclidine, tricyclic antidepressant, buprenorphine, methylenedioxymethamphetamine)
* Use of cannabis products, including CBD, during the past three weeks (determined with urine screen and self-report). Urine drug screen will be performed at each encounter. (Note: Epidiolex is known to sometimes cause a false positive for THC on urine toxicology; drug screen in visit after first CBD administration will not include THC as not to diminish the study blind. Stored urine will be tested for THC after study blind is opened).
* Use of medication altering BOLD response, neurometabolic/glutamatergic levels, and endocrine function, including psychotropic medications (e.g., SSRIs), during the past three months.
* Participation in non-medication-based treatments for anxiety or heightened stress, including cognitive behavioral therapy or other evidence-based treatments, in the past three months.
* Medical or psychiatric contraindications for CBD administration (e.g., history of hypersensitivity to cannabinoids) or any of the ingredients in the product (sesame oil).
* Being pregnant or breastfeeding.
* Not using an appropriate method of contraception such as hormonal contraception (oral hormonal contraceptives, Depo-Provera, Nuva-Ring), intrauterine device (IUD), sterilization, or double barrier method (combination of any two barrier methods used simultaneously, i.e., condom, spermicide, diaphragm).
* Participating in another pharmacotherapeutic trial in the past three months.
* History of impaired renal function or elevated liver enzymes at prescreening. The exclusionary lab values are: 3x normal AST/ALT, 1.5x bilirubin or <30mL/min/1.73m2 eGFR, or QTc>500.
* Participants who have used any medication, dietary supplements (and/or grapefruit juice), or combination of medications and supplements known to alter the metabolism of, or interact with CBD (bupropion, rifampin, barbiturates, phenothiazines, cimetidine, etc.) 14 days prior to and during the duration of the study.
* Any condition that would make study participation unsafe and/or which would prevent adherence to study procedure (e.g., suicidal or homicidal ideation requiring immediate attention, severe inadequately treated mental health condition) as determined by the study clinician and/or PI.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Neural (BOLD) functional response | Day 2
  Measurement of brain activity using the Blood Oxygenation Level Dependent (BOLD) signal Neural (BOLD) functional response to acute stress and network hierarchy in resting state functional connectivity. BOLD response will measure neural activity during stress conditions as compared to rest and control conditions
Neuronal viability indexed by GLX (combined glutamate/glutamine levels) and N-acetylaspartate (NAA) using 1H-MRS. | at day 2
  Concentration of brain chemicals (N-acetylaspartate, Glutamate/Glutamine Levels) as an indicator of brain health measured using non-invasive imaging of magnetic resonance spectroscopy.
Serum Cortisol level | Day 2, Day 3
  The cortisol blood test measures the level of cortisol in the blood. Cortisol is a steroid (glucocorticoid or corticosteroid) hormone produced by the adrenal gland.
Salivary Cortisol level | Day 2, Day 3
  The cortisol saliva test measures the level of cortisol in the saliva. Cortisol is a steroid (glucocorticoid or corticosteroid) hormone produced by the adrenal gland.

SECONDARY OUTCOMES:
Visual analog scale for stress (VASStress) | Day 2, Day 3
  The VASStress consists of a continuous line, usually 10 centimeters long which is converted to a score. Full scale is scored from 0-10, with higher score indicating higher level of stress.
Visual analog scale for anxiety (VASAnxiety) | Day 2, Day 3
  The VASAnxiety consists of a continuous line, usually 10 centimeters long which is converted to a score. Full scale is scored from 0-10, with higher score indicating higher level of anxiety.
Adrenocorticotropic hormone (ACTH) level | Day 2, Day 3
  The ACTH test measures the level of adrenocorticotropic hormone (ACTH) in the blood. ACTH is a hormone released from the pituitary gland at the base of the brain.
Serum noradrenaline level | Day 2, Day 3
  Serum noradrenaline assesses adrenal gland function and the body's response to stress.

CONTACTS AND LOCATIONS:
Overall Officials: Keren Bachi, PhD, Principal Investigator — Ichan School of Medicine
Locations (1):
- Ichan School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared with the National Data Archive of the NIMH per grant requirements.

REFERENCES:
- See also: Prescreen Survey — https://redcap.mountsinai.org/redcap/surveys/?s=M9CWHXECDLTWDHFR